CLINICAL TRIAL: NCT07329933
Title: Effect of Dexamethasone, Dexmedetomidine and Their Combination on Postoperative Gastrointestinal Function Measured by I-FEED Score After Elective Laparoscopic Cholecystectomy Surgery: a Randomized Controlled Trial
Brief Title: Dexamethasone, Dexmedetomidine and Their Combination on Post op. GIT Function Measured by I-FFED Score Post Laparoscopic Cholecystectomy
Acronym: GIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Taghreed Elshahat Sakr, lecturer of anesthesia and icu, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RC.3.11.2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: GIT Function; Cholecystectomy, Laparoscopic; Dexamethasone; Dexmedetomidine; I-FEED Score
MeSH Terms: interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group D (Dexamethasone) (Active Comparator)
  Interventions: Drug: Dexamethasone
- Group X (Dexmedetomidine) (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group DX (Combination) (Active Comparator)
  Interventions: Drug: Dexamethasone and dexmedetomidine
- Group P (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Participants will receive Dexamethasone 8 mg IV + Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia.
  Arms: Group D (Dexamethasone)
Drug: Dexmedetomidine — Participants will receive Dexmedetomidine 0.5 mcg /kg IV + Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia.
  Arms: Group X (Dexmedetomidine)
Drug: Dexamethasone and dexmedetomidine — Participants will receive Dexamethasone 8 mg IV + Dexmedetomidine 0.5 mcg/kg IV+ Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia
  Arms: Group DX (Combination)
Drug: Placebo — Participants will receive Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia
  Arms: Group P (Placebo)

SUMMARY:
The goal of this clinical trial is to learn the effect of Dexamethasone and Dexmedetomidine and Their Combination on Post op. GIT Function Measured by I-FFED Score Post Laparoscopic Cholecystectomy

What medical problems do participants have when taking Dexamethasone and Dexmedetomidine? Researchers will compare Dexamethasone and Dexmedetomidine and Their Combination to a placebo (a look-alike substance that contains no drug) to see the effect on Post op. GIT Function Measured by I-FFED Score Post Laparoscopic Cholecystectomy Participants will receive Dexamethasone 8 mg IV + Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia.

Participants will receive Dexmedetomidine 0.5 mcg /kg IV + Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia.

Participants will receive Dexamethasone 8 mg IV + Dexmedetomidine 0.5 mcg/kg IV+ Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia.

Participants will receive Saline IV (total volume 10 ml) over 10 minutes administered after induction of anesthesia

ELIGIBILITY:
Inclusion Criteria:

- . Age 18-65 years. 2. American Society of Anesthesiologists (ASA) physical status I or II. 3. Scheduled for elective laparoscopic cholecystectomy surgery under general anesthesia.

4. Ability to provide written informed consent

Exclusion Criteria:

* Known allergy or contraindication to any study drug (dexamethasone, dexmedetomidine, or placebo).

  2. Pre-existing gastrointestinal motility disorders (e.g., gastroparesis, inflammatory bowel disease).

  3. Chronic use of opioids, steroids, or antiemetics. 4. History of severe cardiac disease (e.g., high-grade AV block, severe bradycardia).

  5. Uncontrolled diabetes mellitus (HbA1c > 8.0%). 6. Emergency surgery or conversion to open surgery. 7. Pregnancy or breastfeeding. 8. Morbid obesity (BMI >40). 9. Severe hepatic or renal dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The highest I-FEED score | 24 -48 hours post operative
  recorded daily from Postoperative Day (POD) 1 to POD 2. The I FEED score is calculated based on five components: Intake, Feeling nauseated, Emesis, Examination, and Duration of symptoms

SECONDARY OUTCOMES:
Time (hours) to first flatus and first defecation | 24-48 hours post operative
Time to tolerate oral intake. | 24-48 hours postoperative
incidence of POGD (defined as I-FEED score > 2) | 24-48 hours postoperative
postoperative nausea and vomiting (PONV), Incidence and severity | 24-48 hours
• Length of hospital stay (days) from surgery to discharge | 1 week post operative
• Any adverse events related to study drugs | 24-48 hours postoperative
Total rescue opioid consumption | 24-48 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No